CLINICAL TRIAL: NCT02524704
Title: Electrical Impedance Tomography (EIT): A Non-radiating Functional Imaging for Cystic Fibrosis
Brief Title: Electrical Impedance Imaging of Patients With Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: Colorado State University (Other)
Collaborators: Children's Hospital Colorado (Other); University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: ColoradoSU
Record Dates: First submitted 2015-08-07; First posted 2015-08-17 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2016-07

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Electrical Impedance Tomography
MeSH Terms: conditions — Cystic Fibrosis | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Healthy controls: Subjects between the ages of 2 and 21 with healthy lungs. Electrical impedance tomography data will be collected during tidal breathing, during 5 to 10 seconds of breath holding, and during FEV1 and FEF 25-75 spirometry maneuvers for subjects over age 8.
- CF patients scheduled for a CT scan: Subjects with CF between the ages of 2 and 21 who are either clinically indicated for a CT scan of the lungs or are scheduled for a pulmonary CT scan as part of their routine care. Electrical impedance tomography data data will be collected during tidal breathing, during 5 to 10 seconds of breath holding, during forced expiratory volume in 1 second (FEV1) and forced expiratory flow (FEF) 25-75 spirometry maneuvers for subjects over age 8, and immediately before or after pulmonary CT scanning.
  Interventions: Device: CT scan
- CF patients with pulmonary exacerbation: Subjects with CF between the ages of 8 and 21 who are being started on intravenous (IV) antibiotics for a clinically diagnosed pulmonary exacerbation.
  Electrical impedance tomography data data will be collected during tidal breathing, during 5 to 10 seconds of breath holding, during FEV1 and FEF 25-75 spirometry maneuvers upon admission for a pulmonary exacerbation and following 7 to 14 days hospitalized treatment including IV antibiotics. Further data will be collected at the same time with CT scanning if the scan is part of the patient's standard of care.
  Interventions: Device: CT scan

INTERVENTIONS:
Device: CT scan — Applied only when part of the patient's standard care
  Groups: CF patients scheduled for a CT scan; CF patients with pulmonary exacerbation

SUMMARY:
The goal of this feasibility study is to evaluate the ability of Electrical Impedance Tomography (EIT) for providing regional and quantitative information about the extent and nature of bronchial obstruction in patients with cystic fibrosis. It is not being conducted to diagnose, treat, prevent, or cure any kind of disease. In electrical impedance tomography low amplitude, low frequency current is applied on electrodes, and the resulting voltage is measured and used to computed the electrical properties of the interior of the chest as they change in time. The computed properties are used to form an image, which can then be used for monitoring and diagnosis.

DETAILED DESCRIPTION:
The goal of this study is to evaluate the ability of Electrical Impedance Tomography (EIT) hardware and software in patients with cystic fibrosis (CF) for providing regional and quantitative information for identifying regions of obstruction and consolidation, and determine whether these measures will correlate with improvements seen after hospitalized treatment for a pulmonary exacerbation (PE). In particular, EIT will be used to identify regions of obstruction (air trapping) and consolidation comprised of atelectasis and airway occlusion (consequences of mucus plugging) in CF patients, and to determine whether EIT can demonstrate the beneficial effects of antibiotic treatment for CF patients with an acute PE by correlating changes in quantitative EIT measures with clinical measures known to improve following therapy, with patients serving as their own controls. Regional changes in air trapping and consolidation from pre to post treatment as indicated by the EIT images will be calculated, with subjects serving as their own control.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 2 and 21 years (Groups 1 and 2)
* Between the ages of 8 and 21 years (Group 3)
* Healthy lungs (Group 1)
* Clinical diagnosis of cystic fibrosis (Groups 2 and 3)
* Clinically indicated for a pulmonary CT scan or will receive one as part of their routine care (Group 2)
* Receiving IV antibiotics for a clinically diagnosed pulmonary exacerbation (Group 3)

Exclusion Criteria:

* Under age 24 months or over age 21.
* No informed consent
* Known congenital heart disease, arrythmia, or history of heart failure, admission to the intensive care unit, wearing a pacemaker or other surgical implant.
* Pregnant or lactating

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: There are three groups in this study. Group 1 consists of healthy controls between the ages of 2 and 21. Group 2 consists of persons with cystic fibrosis between the ages of 2 and 21 who are either clinically indicated for a pulmonary CT scan or will receive one as part of their routine care. Group 3 consists of persons with cystic fibrosis between the ages of 8 and 21 who are being started on IV antibiotics for a clinically diagnosed pulmonary exacerbation.
  Sampling is by convenience or invitation to volunteer.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2015-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity for identifying air trapping and consolidation | 2 years
  The sensitivity and specificity of EIT for identifying regions of air trapping and consolidation will be assessed using the CT scan as the gold standard

SECONDARY OUTCOMES:
Accuracy of the EIT computed spirometry values | 2 years
  The accuracy of the spirometry measures computed from EIT images will be assessed by comparing to those from the pulmonary function tests
Correlation of EIT derived measures to patient improvement following IV antibiotics | 2 years
  Changes in quantitative EIT measures will be correlated with clinical measures known to improve following therapy, patients serving as their own controls.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Mueller, PhD, Principal Investigator — Colorado State University

REFERENCES:
- [Background] Hamilton SJ, Mueller JL. Direct EIT reconstructions of complex admittivities on a chest-shaped domain in 2-D. IEEE Trans Med Imaging. 2013 Apr;32(4):757-69. doi: 10.1109/TMI.2012.2237389. Epub 2013 Jan 9. PMID 23314771
- [Background] Herrera CN, Vallejo MF, Mueller JL, Lima RG. Direct 2-D reconstructions of conductivity and permittivity from EIT data on a human chest. IEEE Trans Med Imaging. 2015 Jan;34(1):267-74. doi: 10.1109/TMI.2014.2354333. Epub 2014 Sep 4. PMID 25203984